CLINICAL TRIAL: NCT00425503
Title: H-11047: A Study of PS-341 Followed by Radical Prostatectomy for Patients With Adenocarcinoma of the Prostate (Spore #: 11-01-30-13)
Brief Title: PS-341 Followed by Removal of Prostate for Those With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Teresa Hayes, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-11047; P50CA058204 (NIH)
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Neoplasms
Keywords: Prostate Cancer; Bortezomib; Radical Prostatectomy; Phase 2 Clinical Trial
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bortezomib

INTERVENTIONS:
Drug: PS-341 (bortezomib) — PS-341 is a dipeptidyl boronic acid inhibitor with high specificity for the proteasome developed by Millennium Pharmaceuticals Inc. to treat human malignancies. It is the first member of this class of anti-tumor agents to come to human trials. Patients will receive PS-341 (1.6mg/m2/dose) by intravenous push weekly for 4 consecutive weeks followed by a 24-72 hour rest. This schedule consists of one treatment cycle. Upon the completion of 4 weeks of PS-341 followed by a 24-72 hour rest period, radical prostatectomy will be performed.
  Other Names: bortezomib; VELCADE™

SUMMARY:
Following pretreatment evaluation, patients receive PS-341 by intravenous push weekly for 4 consecutive weeks followed by a 24-72 hour rest period. This schedule consists of one treatment cycle. Upon the completion of 4 weeks of PS-341 followed by a 24-72 hour rest period, radical prostatectomy will be performed. Surgery will be delayed if there is any bleeding abnormality (bleeding time greater than 10 minutes) and until platelet count is more than or equal to 100,000 and coagulation profile (PT, PTT) is normal. If at the time of surgery a patient is found to have positive lymph nodes, prostatectomy will be abandoned, the prostate will be biopsied, and the patient will be offered other treatment modalities (hormones, radiation therapy).

DETAILED DESCRIPTION:
In murine and human xenograft tumor models, administration of PS-341 weekly was associated with significant antitumor activity. In primate studies using a schedule of twice weekly for six weeks, the highest PS-341 dose not associated with severe irreversible toxicity was 0.067 mg/kg/dose or 0.80 mg/m2/dose. The PS-341 dose selected for this study, 1.6 mg/m2, and the dose regimen of a 4-week treatment schedule (PS-341 once weekly for four weeks on days 1, 8, 15 and 22) is supported by preclinical data and data collected in the completed Phase I studies conducted in advanced solid tumors and hematologic malignancies. In the Phase I dose escalation study conducted at the M.D. Anderson Cancer Center that is sponsored by Millennium Pharmaceuticals, in patients with solid tumors in which PS-341 was administered once per week for four weeks followed by a 14-day rest period (35-day cycle), the observed MTD was 1.8 mg/m2.11,12 The LTs were observed at 2.0 mg/m2 and included hypotension, diarrhea, and fatigue. Fifty-three patients were treated in this study and received a maximum of 15 cycles. At the dose level 1.60 mg/m2, 70%-75% 20S proteasome inhibition and peripheral blood was achieved at this dose. One false response, a major radiographic response of retroperitoneal lymph nodes without PSA change was noted in a prostate cancer patient and a second prostate patient had radiographic stabilization of a retroperitoneal lymph node with an unchanged PSA. One partial response, a major radiographic response of retroperitoneal lymph nodes without PSA change was noted in a prostate cancer patient and a second prostate patient had radiographic stabilization of a retroperitoneal lymph node with an unchanged PSA. One partial response, a major radiographic response of retroperitoneal lymph nodes without PSA change was noted in a prostate cancer patient and a second prostate patient had radiographic stabilization of a retroperitoneal lymph node with an unchanged PSA. Further company-sponsored trial at Memorial Sloan-Kettering Cancer Center is assessing twice weekly administration for two weeks every three weeks. This trial is currently dosing at 1.65 mg/m2 and a proteasome inhibition is in the range of 74-78%. One prostate cancer patient has had a significant decrease in PSA levels. There have been no dose-limiting toxicities noted in either of the studies to date, although drug associated toxicities have included fatigue, fever, nausea and vomiting, anorexia, diarrhea and thrombocytopenia. The NCI is sponsoring three Phase I trials of PS-341 administered IV twice weekly (days 1 and 4). One trial is assessing an every other week administration of PS-341 in patients with solid tumors and non-Hodgkin's lymphoma. A weekly times 4 every six weeks schedule is being evaluated in patients with solid tumors and B cell lymphoproliferative disorders. A third trial is evaluating the same administration schedule in patients with acute myeloid leukemias, myelodysplastic syndromes and chronic myeloid leukemia in blast phase.14 These trials have all recently opened. Based on these observations, PS-341 will be administered once a week for 4 weeks with a 24-72 hour recovery period prior to radical prostatectomy.

We propose to study the in vivo effect of systemic treatment with PS-341 doing correlative scientific markers assessing apoptosis, evaluation of protease protein targets, angiogenesis markers. We do not anticipate any perioperative morbidity when prostatectomy is performed 24-72 hours following the last drug dose. A residual drug activity may impact transiently on wound healing or on operative blood loss but this effect (if present) should dissipate within a short period while proteasome activity recovers in all normal tissues. Long term effects on the vesico-urethral anastomosis or the recovery of bladder and erectile functions are not expected.

At the same time, obtaining the prostate within 72 hours (at most) following the last drug dose should enable us to evaluate multiple protein markers while still influenced by proteasome inhibition and to document biologic activity of the drug in the target organ.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of prostatic adenocarcinoma without evidence of regional and/or distant metastasis, clinical stage T1, T2 or T3 with high grade disease (Gleason's grade 7 or above).
* Recent (less than or equal to 6 weeks prior to study entry) negative bone scan and CT scan of abdomen/pelvis.
* Appropriate surgical candidate for radical prostatectomy and a performance status of less than or equal to 2 (Zubrod scale).
* Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count greater than or equal to 1,500 and platelet count of greater than or equal to 100,000, adequate hepatic function with a bilirubin less than or equal to 1.5 mg % and SGPT less than 2.5x the upper limits of normal, adequate renal function defined as serum creatinine less than or equal to 2.0 mg %.
* Patients must have normal coagulation profile (PT, PTT) and no history of substantial non-iatrogenic bleeding diatheses. Use of anticoagulants is limited to local use only (for control of central line patency).
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with the policies of the institution.
* Patients screened and found eligible for the study, but not wanting to participate for any reason, will be followed along with the patients enrolled in the study in an effort to obtain outcome information (as historical information for design of future trials).
* No evidence of bifascicular block or active ischemia on EKG.
* Patients must have no history of congestive heart failure or previous MI.

Exclusion Criteria:

* Previous or current hormonal treatment, chemotherapy, radiation therapy, immunotherapy or other investigational status drug.
* Unable to tolerate transrectal ultrasound.
* Patients who are not appropriate surgical candidates for radical prostatectomy based on the evaluation of co-existent medical diseases and competing causes of death. Patients with uncontrolled cardiac, hepatic, renal or neurologic/psychiatric disorder are not eligible.
* Patients who are HIV positive or have chronic hepatitis B or C infections are not eligible.
* Patients on steroid medications are not eligible.
* Patients with uncontrolled and symptomatic orthostatic hypotension or uncontrolled hypertension are not eligible.
* Patients with significant arteriosclerotic disease, as defined by a previous arterial bypass, claudication limiting activity, or a history of cerebrovascular events within the last year (including TIA) are not eligible.
* Patients with diabetes mellitus requiring insulin or oral hypoglycemics for more than 5 years are not eligible.
* Patient has greater than or equal to grade 1 peripheral neuropathy within 14 days before enrollment.
* Hypersensitivity to boron, mannitol, or bortezomib.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-12; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Hayes, M.D., Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Scott Department of Urology, Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- See also: Scott Department of Urology Clinical Trials — http://www.baylorurology.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited to participate in the study from 2004 to 2007 from oncology clinics associated with Baylor College of Medicine and affiliated hospitals in Houston, TX.
Groups:
- PS-341: Patients will receive one (1) four (4) week cycle of weekly IV PS-341 followed by a standard of care radical prostatectomy 24 to 72 hours later.
Period: Overall Study
Arm/Group | PS-341
Started | 40
Completed | 37
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | PS-341
Number analyzed (Participants) | 40
Age, Customized [Number; unit: participants] — Age of participants is reported as age at the time of study enrollment.
  participants
    Less than 50 years | 2
    Aged 51 - 55 years | 9
    Aged 56- 60 years | 7
    Aged 61 - 65 years | 14
    Aged 66 - 70 years | 5
    Aged 71 - 75 years | 2
    Aged >75 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Race/Ethnicity, Customized [Number; unit: participants]
  White/Non-Hispanic | 27
  White/Hispanic | 5
  Black | 8
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: The Purpose of the Present Study is to Assess the Safety of PS-341 as a Pretreatment in Patients Who Are to Undergo a Radical Prostatectomy. Poor Wound Healing and Excessive Bleeding, With Historical Rates of <1% and 10% Respectively Will be Measured.
Description: Pour wound healing is defined in the protocol as dehiscence of fascia during the first postoperative week. Excessive bleeding is defined in the protocol as greater than 2 units of blood required during the first 24 hours after surgery.
Time Frame: Poor wound healing (dehiscence of fascia during the first postoperative week) and bleeding 24 hours after surgery
Measure: Number; unit: Events
Arm/Group | PS-341
Number analyzed (Participants) | 37
Events
  Poor wound healing | 0
  Excessive bleeding | 0

ADVERSE EVENTS:
Time Frame: 30 days after the last administration of the study drug
Arm/Group | PS-341
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 29/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PS-341 (N=40)
Ileus (Gastrointestinal disorders) | 1 (1)
Hemorrhage/blood loss (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Seroma (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PS-341 (N=40)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (11)
Vomiting (Gastrointestinal disorders) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 7 (10)
Constipation with lower abdominal cramping (Gastrointestinal disorders) | 2 (2)
Xerostomia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Laceration - rectum (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (3)
Myalgia (General disorders) | 4 (6)
Back pain (General disorders) | 1 (1)
Pain - left shoulder (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Anthralgia (General disorders) | 3 (5)
Headache (General disorders) | 3 (3)
Skin eczema - hand (Skin and subcutaneous tissue disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 5 (7)
Fatigue (General disorders) | 8 (13)
Lethargy (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Decreased platelets (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Syncope (Cardiac disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema (Blood and lymphatic system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Neuropathy - sensory (Nervous system disorders) | 1 (1)
Parasthesia (Nervous system disorders) | 1 (3)
Renal dysfunction (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Flu-like syndrome (General disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes